CLINICAL TRIAL: NCT06331585
Title: Phase II Trial of Low-dose Radiotherapy (LDRT) Affecting the Tumor Immune Microenvironment (TME) in Oligometastasis, Oligoprogression, and Oligopersistence of Non-small Cell Lung Cancer (NSCLC) After Immunotherapy.
Brief Title: Effect of Low-dose Radiotherapy on Tumor Immune Microenvironment in Oligometastases of NSCLC After Immunotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: work commitments
Sponsor: Hetian District People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KY-2024004
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: Low-dose Radiotherapy; Tumor Microenvironment; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Experimental: LDRT on oligometastasis, oligoprogression, and oligopersistence of NSCLC after immunotherapy
  1. LDRT: Patient undergoes LDRT using a medical linear gas pedal (5Gy/5f)
  2. Biopsy: Collect pathological tissues from oligometastasis, oligoprogression, and oligopersistence of NSCLC after immunotherapy before LDRT (5Gy/5f) and up to 24h after LDRT
  Interventions: Radiation: low dose radiotherapy

INTERVENTIONS:
Radiation: low dose radiotherapy — LDRT (5Gy/5f) of oligometastasis, oligoprogression, and oligopersistence of NSCLC after immunotherapy

SUMMARY:
The purpose of this phase Ⅱ trial was to investigate the effect of low-dose radiotherapy (LDRT) on the tumor immune microenvironment (TME) in oligometastasis, oligoprogression, and oligopersistence of non-small cell lung cancer (NSCLC) after immunotherapy. At least 20 participants will be enrolled in this study. All will take part at Hetian District People's Hospital.

DETAILED DESCRIPTION:
LDRT targeting oligometastases has been shown to enhance anti-tumour immunity by reprogramming the TME, thereby improving the efficacy of immunotherapy. The aim of this study was to collect pathological tissues from oligometastasis, oligoprogression, and oligopersistence of NSCLC after immunotherapy before LDRT (5Gy/5f) and up to 24h after LDRT in order to apply multiplexed fluorescence immunohistochemistry (mIHC) for evaluation of the tumor immune microenvironment. This study will be able to investigate the effect of LDRT on TME in oligometastatic lesions of NSCLC after immunotherapy and assess the efficacy and safety of LDRT.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to take pathologic biopsies of oligometastasis, oligoprogression, or oligopersistence lesions before and up to 24h after LDRT. And be willing and able to provide written informed consent/assent for the trial.
2. Patients with histologically or cytologically confirmed NSCLC.
3. Patient developed oligometastasis, oligoprogression or oligopersistence after standard immunotherapy.
4. Be ≥18 years of age on day of signing informed consent.
5. Be willing to undergo repeat biopsy of tumor lesions according to the study protocol.
6. Patients who have failed the standard therapy, or who are unsuitable for standard treatment, or refuse chemotherapy.
7. At least one measurable lesion according to RECIST 1.1. A lesion that has previously received radiotherapy can be considered a target lesion only if this lesion is clearly progressed after radiotherapy.
8. The target lesions (irradiated lesions) are > 5cm in in diameter
9. ECOG 0-2.
10. Life expectancy of > 3 months.
11. Patients must have normal organ and bone marrow function as defined below: Total bilirubin </= 1.5 x upper limit of normal (ULN). Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Alanine Aminotransferase (ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) <2.5 X institutional upper limit of normal (</= 5 X institutional ULN for subjects with liver metastases) *WBC >/= 3500/uL, ANC >/= 1500/uL *Platelets >/= 90K/ul *Hemoglobin >/= 9g/dL *Creatinine </= 1.5 x ULN, or creatinine clearance ≥ 50 ml/min（Cockcroft-Gault equation）. Coagulation: International Normalized Ratio (INR)≤ 1.5 × ULN, Partial thromboplastin time (PTT) ≤1.5 × ULN; left ventricular ejection fraction (LVEF) >/= 50% and QTcF (Fridericia's formula) ≤ 450ms
12. Patients has recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
13. Wash out period for chemotherapy is more than ≥ 4 weeks, for targeted small molecule therapy ≥ 5 half-lives; palliative radiotherapy must have been completed for at least ≥ 2 weeks, chest radiotherapy must have been completed for at least ≥ 4 weeks, and major surgery must have been completed for ≥ 4 weeks.
14. Subjects with no severe pulmonary ventilation dysfunction, no acute heart failure, and no contraindication to radiotherapy as judged by the radiotherapist. Subjects who agree to receive immunotherapy and radiotherapy treatment.
15. Subjects should agree to use an adequate method of contraception.

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or spinal cord compression, etc.
2. With oncologic emergencies that require immediate treatment
3. EGFR/ALK/ROS-1 mutation or mutation status unknown.
4. Has evidence of interstitial lung disease or active and/or non-infectious pneumonitis (drug-induced pneumonia, radiation-induced pneumonia, etc.) requiring steroid therapy.
5. History of pulmonary fibrosis, pulmonary hypertension, severe irreversible airway obstruction disease
6. Patients with peripheral neuropathy.
7. Significant heart disease or impairment of cardiac function
8. Fluid accumulating in the third space, such as pericardial effusion, pleural effusion and peritoneal effusion that remains uncontrolled by aspiration or other treatment
9. Known allergy to drugs or excipients, known severe allergic reaction to any of the PD-1 monoclonal antibodies
10. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia; treatment with oral or intravenous antibiotics within 2 weeks prior to the start of study treatment; patients receiving prophylactic antibiotic therapy (e.g., to prevent urinary tract infection or exacerbation of COPD) are eligible for this study.
11. Known or suspected active autoimmune disease (congenital or acquired) such as uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. (patients with vitiligo, or resolved childhood asthma may be enrolled; patients with type I diabetes with good insulin control may also be enrolled)
12. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Analysis of the tumor immune microenvironment | 12 months
  mIHC: Multiplex fluorescence immunohistochemical analysis was performed on the collected pathological tissue samples(before LDRT (5Gy/5f) and up to 24h after LDRT) using equipment such as fluorescence microscope and flow cytometer. To reveal the effect of LDRT on the tumor immune microenvironment by detecting the expression of different immune markers.

SECONDARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measurement of Safety and Tolerability of Low Dose Radiotherapy | 48 months
  Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measurement of Safety and Tolerability of Low Dose Radiotherapy
Progression Free Survival (PFS) | 48 months
  Investigator assessed PFS according to RECIST v1.1. Progression free survival is defined as time of enrollment to first evidence of progressive disease up to 48 months after the enrollment
Overall Survival (OS) | 48 months
  OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause up to 48 months after the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Hetian District People's Hospital, Hetian, Xinjiang Uygur Autonomous Region, China

IPD SHARING:
Plan to Share IPD: No